## Official Title: IVY: Intervention for Victimized Youth

NCT Number: NCT06631274 Document Date: October 18, 2024

IRB approved Informed Consent Form

## Block 1

| Click to write the question text |
|------------------------------------------------------|
| I'm not a robot reCAPTCHA Privacy-Terms |
| Interest Survey: Parent |
| Your Name |
| From where are you taking this survey? (City, State) |
| Your phone number |
| Your email address |
| Your home address |
| Child's Name |

O No

Child's grade level Child's school Location of Child's School (City, State) Has your child reported being bullied recently? If enrolled in the program, would your child have access to a tablet or computer with a webcam? A smart phone will not work. O Yes O No If enrolled in the program, would your child have access to a private location for the meeting where there is no one else in the room that could overhear their conversation. Yes

#### Name of Child's School

#### Parent/Guardian Permission

Title of the Study: IVY: An Intervention for Victimized Youth

**Principal Investigator**: Lyndsay Jenkins, Ph.D., NCSP, Licensed Psychologist, Michael and Jean Shahnasarian Endowed Associate Professor, Educational Psychology and Learning Systems.

Your child is being invited to take part in a research study. Please find below information about this research for you to think about before you decide to allow your child to take part. Ask us if you have any questions about this information or the research before you decide to allow your child to take part.

#### **Key Information for You to Consider**

- Statement of the Research Study. Your child is being invited to volunteer to take part in our research study. It is up to you whether your child takes part or not. There will be no penalty or loss of benefits to you or your child if you choose not to have your child take part or decide later to not have them take part.
- **Purpose.** The reason that we are doing this research is to evaluate the effectiveness and relevance of a program that was created to provide support to targets of peer victimization in grades 6-8.
- Duration. Taking part in our program will last eight weeks. Research Activities. Your child will be asked to answer questionnaires and participate in an 8-week small group intervention. Sessions will be held once a week for 45 minutes.
- Risks. The risks or discomforts to your child of taking part in this study include covering sensitive information, such as recalling personal events of peer victimization.
- **Benefits.** As a result of taking part in this research, we think that your child may learn a variety of skills for coping with emotional difficulties and protecting themselves. The goal is to alleviate some of the distress participants may be facing.

## What is this study about?

Researchers at Florida State University are studying interventions for victims of peer victimization. Researchers are interested in finding out whether an intervention they have created is useful for reducing distress associated with peer victimization and teaching skills about how to handle it in the future. Your child is invited to take part in the study because they are a middle school student in Florida who has experienced peer victimization and has expressed distress due to that experience. Your child will participate in a small group (4-8 people) intervention. Their involvement in the study is expected to last 8 weeks.

The study is supported by the National Institutes of Health Grant Number 1R21HD112660-01.

#### What will happen during this research?

If you agree for your child to be in this research, your child's participation will include (1) completing a set of 8 surveys two times (once before and once after the intervention) and (2) participating in an 8 week intervention, which will be held virtually using a HIPAA compliant virtual conference platform (i.e., Zoom). You have the right to inspect these surveys prior to your child's completion of them. Please contact Lyndsay Jenkins for more information.

## What will you do to protect my child's privacy?

The study's results may be published or presented, but no information that may identify your child will ever be provided or released. We will take steps to protect your child's privacy and confidentiality. These steps include using ID numbers instead of names, storing information on a password-protected server that only research staff has access to, and collecting survey data on a password-protected site (i.e., Qualtrics). Despite taking steps to protect your child's privacy or the confidentiality of their identifiable information, we cannot guarantee that their privacy or confidentiality will be protected. For example, if your child tells us something that makes us believe that they or others have been or may be physically harmed, we may need to report that information to the appropriate agencies.

Individuals and organizations responsible for conducting or monitoring this research may be permitted access to and to inspect the research records. This includes the Florida State University Institutional Review Board (FSU IRB), which reviewed this study.

If identifiers are removed from your child's identifiable private information that is collected during this research, that de-identified information could be used for future research studies or distributed to another investigator for future research studies without your additional informed consent.

#### What are the risks of harm or discomfort associated with this research?

Given the sensitive nature of the IVY intervention, it is likely that the participants may feel distressed or uncomfortable when discussing or recalling events when they were the target of peer victimization. Sharing their victimization stories is encouraged during one session, but it will not be required. There is a risk that group members may share experiences or events that could be considered harassment or abuse. To alleviate any distress caused by the intervention, group leaders will be available to individuals after the sessions. In addition to the risks of these harms or discomforts, this research may have risks of harm or discomfort that are unknown at this time. If, in the future, we become aware of any additional harm or discomfort that may affect your child, we will tell you.

#### How might my child benefit from this research?

Personal direct benefits your child may get from this study include (1) fewer feelings of distress (e.g., sadness, anxiousness, worry), (2) support from peers who have experienced the same thing as them, and (3) skills for handling future victimization and distress. These are the goals of the IVY program.

## What is the compensation for the research?

Participants will receive a gift card if they complete the pre-test, 8-week intervention, and post-test. They must be present for at least 6 of the 8 sessions. Partial completion will not be compensated, nor will early withdrawal from the study.

## What will happen if I choose not to participate?

It is your choice to have your child participate in this research. Participation is voluntary.

## Is my child's participation voluntary, and can they withdraw?

Having your child take part in this research study is your decision. Your child's participation in this study is voluntary. Your child does not have to take part in this study, but if your child does, they may stop at any time. Your decision to have your child participate will not affect your or your child's relationship with these researchers or FSU.

Your child will not receive compensation if they withdraw early. If they withdraw from the study, the data collected to the point of withdrawal will be deleted.

#### Can my child be removed from the research without my OK?

We may remove your child from the research study without your approval. Reasons we would do this include if your child is being disrespectful to other participants in the group or if they become too distressed to continue in a healthy manner.

#### Who do I talk to if I have questions?

If you have questions, concerns, or have experienced a research-related injury, contact the research team at:

Lyndsay Jenkins, Ph.D.

850-644-9445

Injenkins@fsu.edu

The Florida State University Institutional Review Board ("IRB") is overseeing this research. The FSU IRB is a group of people who perform official independent research reviews before studies begin to ensure that participants' rights and welfare are protected. If you have questions about your rights or wish to speak with someone other than the research team, you may contact:

Florida State University IRB 2010 Levy Drive, Suite 276 Tallahassee, Florida 32306 850-644-7900 humansubjects@fsu.edu

#### STATEMENT OF CONSENT

I have read and considered the information presented in this form. I confirm that I understand the purpose of the research and the study procedures. I understand that I may ask questions at any time and can withdraw my child's participation without prejudice. I have read this consent form. My signature below indicates my willingness to allow my child to participate in this study. I consent to my child participating in this study.

# SIGN HERE

| × | |
|---|---|
| clear | |
| If your child participates in the program, the university researched that we receive consent from both parents, if there is a second | · |
| Yes, there is a second parent to provide consent No, there is not a second parent to provide consent | |
| Please provide contact information for Parent #2. We will conta<br>permission. | act them to get their |
| Typed Name of Parent/Guardian #2 | |
| Parent/Guardian #2 Email Address | |
| Parent/Guardian #2 Phone Number | |
| Powered by Qualtrics | |

Qualtrics Survey Software

10/18/24, 4:25 PM